CLINICAL TRIAL: NCT03660020
Title: Effect of Hyalorounidase on the Spread of Local Anaesthetics in Erector Spinae Plane Block
Brief Title: Ultrasound Guided Erector Spinae Plane Block in Breast Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rasha Hamed, clinical professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NBBL
Record Dates: First submitted 2018-07-20; First posted 2018-09-06 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthetics, Local; Hyaluronoglucosaminidase

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- local anaesthetic group (Sham Comparator)
  Interventions: Drug: Local anesthetic
- hyalorounidase group (Active Comparator)
  Interventions: Drug: Hyaluronidase

INTERVENTIONS:
Drug: Local anesthetic — ultrasound guided erector spine plane block (ESP) will be done in patients under going mastectomy with local anaesthetics only
  Arms: local anaesthetic group
Drug: Hyaluronidase — hyaluronidase will be added to ultrasound guided erector spine plane block (ESP) will be done in patients under going mastectomy
  Arms: hyalorounidase group

SUMMARY:
hyalorounidase will be added to local anaesthetics in patients undergoing mastectomy and effect on local anaesthetic spread will be studied under floroscope

DETAILED DESCRIPTION:
two groups will be enrolled the control group will receive local anaethetic only and the spread will be observed by floroscope. the seconed group, hyaloronidase will be added to local anaesthetics and the spread will be studied under image.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. ASA I, II, III
3. Elective surgery

Exclusion Criteria:

1. Patient refusal
2. Infection at injection site
3. Allergy to the given drugs

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-05-19 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
degree of local anaesthetics spread after injection in both group | 10 minutes after block
  spread of local anaesthics will be examined under floroscopic guide

CONTACTS AND LOCATIONS:
Overall Officials: saeid elsawy, Study Chair — Assiut University
Locations (1):
- Assiut university, Asyut, Egypt